CLINICAL TRIAL: NCT00484848
Title: Functional Evaluation of Conventional Venous Access Port (Celsite®) Versus Venous Access Port With Tangential Outlet (Vortex®) : a Prospective Randomized Pilot Study
Brief Title: Functional Evaluation of Two Types of Totally Implanted Venous Ports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: RITA Medical Systems (Industry); B. Braun Medical SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SM007
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Hematologic Disease
Keywords: oncology, medical; implantable catheter; vascular access ports; persistent withdrawal occlusion; Vortex®; Celsite®; Vacutainer®; venous cut-down
MeSH Terms: conditions — Hematologic Diseases; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vortex port and Celsite port

SUMMARY:
Totally implanted venous access ports allow a safe delivery of medication, mainly chemotherapy, but are also used for blood sampling. This last procedure is not always successful, as it appeared from a nurse's survey in different hospitals in Flanders, including the University Hospitals in Leuven, Belgium. In 3 to 29 percent of the attempts, blood withdrawal is impaired or not possible, as an intermittent or permanent fact. This is in line with international literature data where difficulty in blood draw was noted in 6 to 26% of port accessions. Partial or total occlusion leads to discomfort for the patient, delay in therapy, higher costs and extra nursing time.

A new port system with a tangential outlet (Vortex port) was designed and according to the manufacturer, this shape will allow to cleanse the entire reservoir of the port more efficiently and avoid the formation of precipitates of medication or blood that could lead to an obstruction of the device. These precipitates are also regarded as a potential risk factor for infection.

However, only one previously published small randomised study addressed the value of the Vortex port when compared to conventional access devices: Stevens et al. were able to show a reduction in obstruction incidence from 26% to 7% with the use of the Vortex port. The incidence of blood withdrawal problems in our experience with conventional ports in University hospitals Leuven was 8% thus lower than that reported by Stevens, but this remains the most frequent problem faced by care providers and patients.

With this study, the investigators aim to compare the performance of the tangential outlet ports and that of a "conventional" port in order to assess an eventual functional difference.

ELIGIBILITY:
Inclusion Criteria:

* request of a standard size totally implanted venous port
* patent superior vena cava
* normal clotting tests (PT>40% and platelet count >40000/mm3)

Exclusion Criteria:

* unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the difference in difficulty in blood drawing between the 2 types of ports when accessing the port under identical maintenance procedure according to the guidelines in the University Hospitals Leuven. | up to a maximum of 6 months after insertion
Evaluation of the difference in one-way or bidirectional occlusion incidence between these 2 types of ports, when accessing the port under identical maintenance procedure according to the guidelines in the University Hospitals Leuven. | up to a maximum of 6 months after insertion
Evaluation of the difference in filling time for blood sampling between these 2 types of ports when using a standard 10 ml vacuum blood tube and a 19 G Gripper® needle. | immediately after insertion and up to a maximum of 6 months afterwards

SECONDARY OUTCOMES:
Evaluation of the ease of use (ease of access) between these 2 types of ports when accessing the port. | up to a maximum of 6 months after insertion

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite Stas, MD PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Stevens B, Barton SE, Brechbill M, Moenter S, Piel AL, Shankle D. A Randomized, Prospective Trial of Conventional Vascular Ports Vs.the Vortex
- [Background] Lamont JP, McCarty TM, Stephens JS, Smith BA, Carlo J, Livingston S, Kuhn JA. A randomized trial of valved vs nonvalved implantable ports for vascular access. Proc (Bayl Univ Med Cent). 2003 Oct;16(4):384-7. doi: 10.1080/08998280.2003.11927932. PMID 16278752
- [Result] Goossens GA, Verbeeck G, Moons P, Sermeus W, De Wever I, Stas M. Functional evaluation of conventional 'Celsite' venous ports versus 'Vortex' ports with a tangential outlet: a prospective randomised pilot study. Support Care Cancer. 2008 Dec;16(12):1367-74. doi: 10.1007/s00520-008-0436-y. Epub 2008 Apr 15. PMID 18414904